CLINICAL TRIAL: NCT04155931
Title: The Effect of Intraoperative Body Temperature on Postoperative Nausea and Vomiting in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, İsmail SÜMER, MD, Principal Investigator, Bezmialem Vakif University
Other Study IDs: İsmail01
Record Dates: First submitted 2019-10-30; First posted 2019-11-07 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Perioperative Body Temperature; Postoperative Nausea and Vomiting
Keywords: perioperative body tempreture; hypothermia; PONV; Postoperative nausea and vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Hypothermia | interventions — Body Temperature

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- body temperature measurement: The investigators planned to perform prospectively in 80 children with ASA I according to the American Society of Anesthesia (ASA) Anesthesia Risk Scale between 6 months and 7 years of age in both sexes who underwent inguinal hernia, undescended testes and hydrocele surgery
  Interventions: Other: body temperature measurement

INTERVENTIONS:
Other: body temperature measurement — Postoperative analgesic and antiemetic requirements, nausea and vomiting were observed in the recovery room at 6, 12 and 24 hours

SUMMARY:
The aim of our study was to investigate the effects of changes in body temperature in the perioperative period on postoperative nausea and vomiting.

DETAILED DESCRIPTION:
Undesirable hypothermia is that the perioperative body temperature is below 36 ° C. Perioperative heat loss is higher in pediatric patients than in adult patients. One of the most common side effects of general anesthesia is nausea and vomiting. The aim of our study was to investigate the effects of changes in body temperature in the perioperative period on postoperative nausea and vomiting.We planned to perform prospectively in 80 children with ASA I according to the American Society of Anesthesia (ASA) Anesthesia Risk Scale between 6 months and 7 years of age in both sexes who underwent inguinal hernia, undescended testes and hydrocele surgery. In all patients, heating blanket was placed on the operation table and standard heat was used. After the placement of the LMA, a nasopharyngeal heat probe was placed for central body temperature measurement and monitored throughout the operation. Mean arterial pressure, heart rate and body temperature were recorded. Demographic data, type of operation, duration of operation and intraoperative fentanyl requirement of all cases were recorded. Analgesic and antiemetic requirements, presence of nausea and vomiting (according to numerical sequence scale) were recorded in the recovery room at 6, 12 and 24 hours postoperatively

ELIGIBILITY:
Inclusion Criteria:

* ASA1 group
* Aged 6 months to 7 years
* lower abdominal and urological surgery

Exclusion Criteria:

* Upper abdominal surgery
* ASA 2-3 group
* postoperative nausea and vomiting history

Ages: 6 Months to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: ASA1 group, 80 children, both sexes, aged 6 months to 7 years
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
hypothermia | intraoperative
  Perioperative body temperature below 36 ° C is defined as unwanted hypothermia. It may cause postoperative neusea and vomiting.
Postoperative Nausea and vomiting | Postoperative 24 hours
  Postoperative analgesic and antiemetic requirements, nausea and vomiting were observed in the recovery room at 6, 12 and 24 hours.The investigators use numerical scale for posteoprative nausea and vomiting. 0-no nausea and vomiting, 1-nausea yes, vomiting no, 2- only 1 episode of vomiting and score3 is multiple vomiting episodes. if score is 1 or more than 1 we apllied antiemetics.

SECONDARY OUTCOMES:
Postoperative Pain | Postoperative 24 Hours
  Postoperative analgesic and antiemetic requirements, nausea and vomiting were observed in the recovery room at 6, 12 and 24 hours. The investigators use pediatric objective pain scale.

CONTACTS AND LOCATIONS:
Overall Officials: İsmail Sümer, MD, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided